CLINICAL TRIAL: NCT02687178
Title: Efficacy and Safety of Canrenone as Add-on in Patients With Essential Hypertension-Italy (ESCAPE-IT)
Brief Title: Canrenone as Add-on in Patients With Essential Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PhD, FESC, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-023606-13
Record Dates: First submitted 2016-02-17; First posted 2016-02-22 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canrenone 50 mg (Active Comparator): Caucasian patients affected by uncomplicated, essential hypertension, not well controlled by concomitant administration of ACE-I or ARBs and diuretics at the maximum dosage.
  Interventions: Drug: Canrenone 50 vs canrenone 100 mg
- Canrenone 100 mg (Active Comparator): Caucasian patients affected by uncomplicated, essential hypertension, not well controlled by concomitant administration of ACE-I or ARBs and diuretics at the maximum dosage.
  Interventions: Drug: Canrenone 50 vs canrenone 100 mg

INTERVENTIONS:
Drug: Canrenone 50 vs canrenone 100 mg

SUMMARY:
To evaluate the efficacy on blood pressure reduction, safety and tolerability of two different dosages of canrenone as add-on therapy in patients already treated with Angiotensin Converting-Enzyme Inhibitors (ACE-I) or Angiotensin II Receptor Blockers (ARBs) and diuretics at the maximum dosage.

DETAILED DESCRIPTION:
To evaluate the efficacy on blood pressure reduction, safety and tolerability of two different dosages of canrenone as add-on therapy in patients already treated with Angiotensin Converting-Enzyme Inhibitors (ACE-I) or Angiotensin II Receptor Blockers (ARBs) and diuretics at the maximum dosage.

In this multi-centre, phase IV, randomized, controlled, open-label, parallel groups trial, 180 Caucasian patients affected by uncomplicated, essential hypertension, not well controlled by concomitant administration of ACE-I or ARBs and diuretics at the maximum dosage will be enrolled.

At baseline patients will be randomized to canrenone, 50 mg, or canrenone 100 mg once a day, in addition to their current therapy, for three months.

At the baseline, and after 3 months will be evaluated: systolic (SBP) and diastolic blood pressure (DBP), pulse pressure (PP), heart rate, fasting plasma glucose (FPG), homeostasis model assessment insulin (HOMA-index), total cholesterol, HDL-cholesterol, triglycerides, LDL-cholesterol, sodium, potassium, calcium, magnesium, uric acid, estimated glomerular filtration rate (eGFR), plasmatic urea, brain natriuretic peptide (BNP), aldosterone, and galectin-3.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian patients affected by uncomplicated, essential hypertension, not well controlled by concomitant administration of ACE-I or ARBs and diuretics at the maximum dosage.

Exclusion Criteria:

* diabetes mellitus
* secondary hypertension
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-10; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Systolic (SBP) and Diastolic blood pressure reduction | 3 months

REFERENCES:
- [Derived] Derosa G, Maffioli P, D'Avino M, Sala C, Mugellini A, Vulpis V, Felis S, Guasti L, Sarzani R, Bestetti A, Vanasia M, Gaudio G; ESCAPE-IT Trial Investigators group. Efficacy and safety of two dosages of canrenone as add-on therapy in hypertensive patients taking ace-inhibitors or angiotensin II receptor blockers and hydrochlorothiazide at maximum dosage in a randomized clinical trial: The ESCAPE-IT trial. Cardiovasc Ther. 2017 Feb;35(1):47-54. doi: 10.1111/1755-5922.12235. PMID 27860389